CLINICAL TRIAL: NCT05685875
Title: Malaria, Diabetes and Metabolic Syndrome: Investigating the Double Burden of Diseases in Cameroon
Brief Title: Association of Diabetes and Metabolic Syndrome With Severe Malaria in Cameroon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Dschang (Other)
Responsible Party: Principal Investigator, Katja Wyss, prinicpal investigator, Karolinska Institutet
Other Study IDs: 2022-05379-01; 2020-05494 (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2022-11-11; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Metabolic Syndrome; Severe Malaria; Malaria,Falciparum
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Metabolic Syndrome; Malaria; Malaria, Falciparum | interventions — Adiposity; ANAPC16 protein, human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples for biochemistry analyses, malaria detection and Ag/serology (HIV) test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diabetes — Diabetes and metabolic syndrome defined using criteria by IDF. Obesity defined as BMI>=30
  Other Names: obesity; metabolic syndrome

SUMMARY:
The aim of this study is to investigate if diabetes, obesity and metabolic syndrome affects disease presentation and severity of malaria in adults in a hospital setting in Cameroon.

DETAILED DESCRIPTION:
Malaria is a major global health problem affecting approximately 241 million people and causing more than 600 thousand deaths, according to the latest WHO estimates. In parallel non-communicable life style diseases increase globally, also in malaria-endemic areas. Surprisingly few studies have investigated possible associations between malaria and non-communicable diseases. Higher prevalence of asymptomatic malaria infection has been shown among individuals with type 2 diabetes in Ghana and the risk of malaria increased with poor glucose control. In a recent study on more than 900 adults with P. falciparum malaria in Sweden, comorbidities and especially diabetes, metabolic syndrome and obesity were associated with a 3-5 times increased risk of severe malaria . Interestingly, these associations were apparent also in African immigrants, a group otherwise recognized to be at reduced risk of severe malaria due to pre-existing immunity. Altered metabolism and chronic inflammatory state in individuals with obesity and diabetes might affect severe progression of malaria. Moreover, poor antibody responses have been observed in obese individuals vaccinated against viral and bacterial infections; and impaired antibody mediated immunity might also affect the risk of malaria.

The overall aim of this project is to investigate whether diabetes, obesity and the metabolic syndrome affects the risk of severe malaria in an endemic setting.

The study will be performed at the District Hospital Dschang and the Bafoussam Regional Hospital in Western Cameroon. Adults diagnosed with malaria at the two hospitals, both at the outpatient clinic and admitted to the hospital wards, will be invited to participate in the study. Informed consent is needed for inclusion. The participants will be clinically evaluated for diabetes and the metabolic syndrome according to International Diabetes Federation (IDF) criteria. In addition to lab parameters below, weight and height will be measured for body mass index (BMI). Severe malaria will be defined according to WHO criteria.

Malaria species and parasite density will be assessed by microscopy of blood films stained with Giemsa. Clinical chemistry will include a fasting plasma glucose, glycated haemoglobin (HBA1c), lipids, erythrocyte sedimentation rate (ESR), liver enzymes, bilirubin, creatinine and haemoglobinopathies such as sickle cell will be assessed. HIV test will be offered to all patients. For patients admitted to hospital, fasting plasma glucose, parasitaemia and insulin levels will be measured on a daily basis. Venous EDTA blood sample will be collected at admission and stored frozen as plasma and packed cells for later PCR confirmation.

ELIGIBILITY:
Inclusion Criteria:

* Adults 20 years and above
* Diagnosed with malaria (all Plasmodium species, confirmed by microscopy)
* Have given consent to participate in the study

Exclusion Criteria:

* Children/youths <20 years

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults, >=20 years diagnosed with malaria (all Plasmodium species), will be recruited prospectively at both the outpatient department (OD), emergency department (ED) and hospital wards in Dschang and Bafoussam hospital. The malaria diagnosis can initially be by rapid test but should be confirmed by microscopy (for sepcies determination and parasite count). Patients will be invited to participate in the study after they return from laboratory investigations following routine consultation at the ED/OD if they have a positive malaria result.
  Participant recruitment will be conducted daily during normal work hours until the estimated study sample is attained. Patients that have seeked health care outside office hours and been admitted for malaria will be recruited the following day.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Severe malaria | 1 year
  P falciparum or other malaria species identified by microscopy and one or more criteria for severe malaria according to WHO 2015 definition.

SECONDARY OUTCOMES:
Malaria requiring in-patient care | 1 year
  Patients with confirmed malaria admitted to hospital
Cerebral malaria | 1 year
  Confirmed malaria and Glasgow Coma Scale <11
Severe malaria with kidney failure | 1 year
  Confirmed malaria and Creatinine >265

CONTACTS AND LOCATIONS:
Overall Officials: Anna Färnert, Prof, Study Director — Karolinska Institutet
Locations (2):
- Cameroon (2):
  - Dschang Hospital, Dschang, West Cameroon
  - Bafoussam Regional Hospital, Bafoussam, West Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wyss K, Wangdahl A, Vesterlund M, Hammar U, Dashti S, Naucler P, Farnert A. Obesity and Diabetes as Risk Factors for Severe Plasmodium falciparum Malaria: Results From a Swedish Nationwide Study. Clin Infect Dis. 2017 Sep 15;65(6):949-958. doi: 10.1093/cid/cix437. PMID 28510633
- [Background] Danquah I, Bedu-Addo G, Mockenhaupt FP. Type 2 diabetes mellitus and increased risk for malaria infection. Emerg Infect Dis. 2010 Oct;16(10):1601-4. doi: 10.3201/eid1610.100399. PMID 20875289
- [Background] Sun H, Saeedi P, Karuranga S, Pinkepank M, Ogurtsova K, Duncan BB, Stein C, Basit A, Chan JCN, Mbanya JC, Pavkov ME, Ramachandaran A, Wild SH, James S, Herman WH, Zhang P, Bommer C, Kuo S, Boyko EJ, Magliano DJ. IDF Diabetes Atlas: Global, regional and country-level diabetes prevalence estimates for 2021 and projections for 2045. Diabetes Res Clin Pract. 2022 Jan;183:109119. doi: 10.1016/j.diabres.2021.109119. Epub 2021 Dec 6. PMID 34879977
- [Background] Guidelines for the Treatment of Malaria. 3rd edition. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK294440/ PMID 26020088
- [Background] Alberti KG, Zimmet P, Shaw J. Metabolic syndrome--a new world-wide definition. A Consensus Statement from the International Diabetes Federation. Diabet Med. 2006 May;23(5):469-80. doi: 10.1111/j.1464-5491.2006.01858.x. PMID 16681555